CLINICAL TRIAL: NCT04947930
Title: Fecal Metagenomics and Metabolomics Analyses to Identify Potential Screening Biomarkers for Colorectal Polyps and Cancer in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ping Lan, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2021SYSUMMS
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer; Colorectal Polyp; Mass Screening; Gastrointestinal Microbiome
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many previous studies had revealed that gastrointestinal microbiome is changed compositionally and ecologically in patients with colorectal cancer comparing with healthy population. These finding provide us with a new sight to take advantage of gut microbiota. The current study aims to explore new potential biomarkers for early screening and prognostic prediction of colorectal cancer and colorectal polyps by analyzing metagenomics and metabolomics of gut microbiota.

DETAILED DESCRIPTION:
Patients who come to the Sixth Affiliated Hospital, Sun Yat-sen University for medical purposes will be invited to participate in the study. Participants will be asked to collect two stool samples. One stool sample will be used for metagenomic sequencing and the other will be used to extract metabolomics data. Meanwhile, participants will be asked to complete a questionnaire about lifestyle and diet habits with the assistance of a well-trained nurse.

We will delineate the community and metabolites differences in the gut microbiota between colorectal cancer patients and healthy populations by comparing cases with controls. Considering the different gut microbiota profiles among different populations caused by varied diet habits and lifestyles, the current study will try to describe the microbiota profiles in the Chinese population. Besides, we will explore new potential biomarkers for early screening and prognostic prediction which is suitable to Chinese populations. Moreover, we will attempt to find out the interactions between diet and microbiota through a comprehensive analysis of the questionnaire and the collected results.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 80 years old.
2. Participants who had been diagnosed with colorectal cancer or advanced colorectal polyps for the first time according to pathology results.
3. Participants who had signed informed consent.
4. Participants must have the ability to complete the questionnaires of the study.

Exclusion Criteria:

1. Participants who had a positive personal history of colorectal polyps.
2. Participants who had a positive personal history of colorectal cancer.
3. Participants who had a positive personal history of other gastrointestinal diseases, such as inflammatory bowel disease， intestinal tuberculosis, or irritable bowel syndrome.
4. Participants who had undergone a colonoscopy or other procedure requiring bowel preparation in the last two months.
5. Participants who had been hospitalized for any reason in the last two months.
6. Participants who had consumed antibiotics for any reason in the last three months.
7. Participants who had consumed prebiotic supplements regularly in the last year.
8. Participants who had other physical conditions that didn't suitable to participate in the study, such as severe cardiovascular diseases, serious mental illness, or pregnant status.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled in the Six Affiliated Hospital, Sun Yat-sen University (Guangzhou, China)，which is one of the largest gastrointestinal specialized medical centers in South China.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the screening tool generated from fecal metagenomics and metabolomics data. | 12months

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lan, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China